CLINICAL TRIAL: NCT03083444
Title: Early P Gingivalis Oral Infection and Ultrasound Detection of Intimamedia Thickening in Radial Arteries of Young Children
Brief Title: P Gingivalis Oral Infection, Intimamedia Thickening in Infants, Atherosclerosis
Status: Withdrawn | Type: Observational
Why Stopped: Grant not funded so clinical trial not started.
Sponsor: Creighton University (Other)
Responsible Party: Principal Investigator, Douglas K Benn DDS, PhD, Professor, Creighton University
Other Study IDs: 925229-1
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Tooth Eruption, Atherosclerosis
MeSH Terms: conditions — Exanthema; Atherosclerosis | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound — Measurement of thickness of radial artery wall thickness by ultrasound

SUMMARY:
To determine if there is an association between Porphyromonas gingivalis infection of dental gingiva during primary tooth eruption and thickening of the radial artery intimamedial layers. Thickening of these layers in infants could be a promoting factor for later development of atherosclerosis.

DETAILED DESCRIPTION:
Specific Aim 1. To determine the presence of Pg in the mouth of edentulous pre-eruption and then teething infants.

Over a 9-month period 15 normal babies will be recruited for a prospective pilot study from Creighton University students. Cotton swabs of the tongue mucosa and dental plaque will be made to detect the presence of Pg by DNA analysis.

Specific Aim 2. To determine the daily temperature of infants. Daily child temperatures will be recorded by the parent. Specific Aim 3. To measure the thickness of the radial artery using a 50 MHz ultrasound probe.

A 50 MHz ultrasound scan will be made by a trained dental hygienist of the left radial artery at an initial visit and at 3-monthly intervals to measure IMT.

ELIGIBILITY:
Inclusion Criteria:

* Pre-primary tooth eruption infants in the range of 4-8 months -

Exclusion Criteria:

* No erupted teeth. No diabetes, obesity, chronic inflammatory disorders, hyperlipidemia, -

Ages: 4 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants 4- 24 months of age.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-04-15 (Estimated); Primary Completion 2018-11-30 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
Arterial wall thickness | 9 months
  Increase in thickness of intimamedia layers

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Benn, DDS PhD, Principal Investigator — Creighton University
Locations (1):
- Creighton University School of Dentistry, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No